CLINICAL TRIAL: NCT05778721
Title: Psychiatric Co-morbidities (Seasonal Affective Disorder and Bipolar Disorder) and Socio-demographic Characteristics in Patients With Idiopathic Hypersomnia: Quantitative Study Following 48-hour Polysomnographic Recordings.
Brief Title: Psychiatric Co-morbidities and Socio-demographic Characteristics in Patients With Idiopathic Hypersomnia
Acronym: HYPERSOMNPSY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/22/0127
Record Dates: First submitted 2022-08-18; First posted 2023-03-21 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Idiopathic Hypersomnia; Mood Disorder; Bipolar Disorder
Keywords: demographic characteristic; psychiatric morbidity
MeSH Terms: conditions — Idiopathic Hypersomnia; Mood Disorders; Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- adult patients with a diagnosis of idiopathic hypersomnia: adult patients with a diagnosis of idiopathic hypersomnia according to the International Classification of Sleep Disorders (ICSD 3) criteria and the performance of a 48-hour polysomnography at the Sleep Laboratory, between 2004 and today.
  Interventions: Other: respond to questionnaires by telephone

INTERVENTIONS:
Other: respond to questionnaires by telephone — Seasonal Pattern Assessment Questionnaire (SPAQ) questionnaires and Sachs bipolarity index and Idiopathic Hypersomnia (IH) severity score

SUMMARY:
This is a study of only patients with idiopathic hypersomnia. It is a rare and still poorly understood pathology. In clinical practice, we have found that the treatment and care offered were not always effective. The idea of this study to improve knowledge of this pathology by studying the demographic characteristics of patients and other co-morbidities, in particular psychiatric patients, to see if we can identify common factor to our patients and useful in their medical care. The main objective of this research is to allow a quantitative study of the demographic and psychiatric characteristics of patients with idiopathic hypersomnia.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with a diagnosis of idiopathic hypersomnia according to the ICSD 3 criteria and the performance of a 48-hour polysomnography at the Sleep Laboratory, between 2004 and today.

Exclusion Criteria:

* minors persons and under legal protection persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with idiopathic hypersomnia
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-06-16 (Estimated); Study Completion 2024-06-16 (Estimated)

PRIMARY OUTCOMES:
demographic characteristics | day 1
  SPAQ questionnaires
psychiatric characteristics | day 1
  SACHS bipolarity index

CONTACTS AND LOCATIONS:
Overall Officials: Rachel DEBS, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Chu Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided